CLINICAL TRIAL: NCT04782947
Title: Epidural Stimulation and Resistance Training for Overground Locomotion After Spinal Cord Injury
Brief Title: Epidural Stimulation and Resistance Training After SCI
Acronym: REST-SCI
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Collaborators: Central Virginia VA Health Care System (Unknown)
Responsible Party: Principal Investigator, Ashraf S. Gorgey, Director of SCI Research, Virginia Commonwealth University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SC190107
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
Keywords: neuromodulation; epidural simulation; exoskeletal assisted walking; resistance training; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- EAW+ES+RT (Experimental): The exoskeletal assisted walking with epidural simulation and resistance training (EAW+ES+RT) group will undergo 6 months of supervised EAW +ES (3X per week) followed by additional 6 months of EAW+ES (3X per week) and progressive RT twice weekly (2X per week). In the EAW+ES+RT group, RT will be administered for 12 weeks using an open kinematic chain approach of applying surface NMES and ankle weights followed by 12 weeks twice weekly of gradually using the implanted ES to perform sit-to-stand approach (i.e. using their body weights to load the exercising muscles in a closed kinematic fashion).
  Interventions: Device: Exoskeletal assisted walking; Device: Epidural Stimulation; Procedure: Resistance Training
- EAW+ delayed-ES +no-RT (Experimental): The control exoskeletal assisted walking with delayed epidural simulation and without resistance training (EAW+ delayed-ES +no-RT) group will enroll in 6 months of EAW without ES (3X per week) and then this will be followed by additional 6 months (3x per week) of EAW+ES (i.e., delayed entry approach) without conducting RT and will perform either passive movement of passive stretching (2X per week).
  Interventions: Device: Exoskeletal assisted walking; Device: delayed-ES; Procedure: no-Resistance training

INTERVENTIONS:
Device: Exoskeletal assisted walking — Exoskeletal assisted walking includes the use of robotic suit to train participant to walk with different level of assistance.
  Other Names: EAW
Device: Epidural Stimulation — lumbo-sacral epidural simulation at the beginning of the study.
  Other Names: ES
  Arms: EAW+ES+RT
Procedure: Resistance Training — Using two forms of resistance training to increase muscle size. The first form includes seated leg extension exercise for 12 weeks followed by a second form that includes sit-to-stand exercise using participant's body weight.
  Other Names: RT
  Arms: EAW+ES+RT
Device: delayed-ES — lumbo-sacral epidural simulation starting 6 months after the beginning of the study.
  Arms: EAW+ delayed-ES +no-RT
Procedure: no-Resistance training — The participants will perform 24 weeks of passive movement or passive stretching from seated position.
  Other Names: no-RT
  Arms: EAW+ delayed-ES +no-RT

SUMMARY:
Spinal cord injury (SCI) is a devastating health problem for tens of thousands of military personnel, Veterans and civilians annually. Many persons with SCI must use a wheelchair for their entire life. A new scientific breakthrough called "lumbosacral epidural stimulation" or "ES" can help people with SCI to stand, step and even walk again. At present, for ES to work, people must train with a specialized treadmill that requires several other qualified personnel to train them, which makes it hard for many people with SCI to benefit from this technology. On the other hand, there are wearable "robot suits" that can be used with ES, which would make it easier to use. Our research team has already used this "ES Robot Suit" for 3 months in one person with tetraplegia and showed remarkable improvements in motor control. Furthermore, the investigators are aiming to enhance overground motor recovery by adding 6 months of resistance training (RT). The addition of RT will likely to enhance muscle quality as indicated by increasing lean mass, peak torque and increase sensory flux to the central nervous system. Other additional benefits may include improvement in cardiovascular profile and bladder functions. The specific objectives of the current proposal are to compare the impact of EAW+ES following improving lower extremity muscle quality compared to those who will only undergo EAW+ ES without conducting RT on motor recovery, cardio-metabolic health and bladder control in persons with complete SCI. At the conclusion of the current proposal, the work will be readily available for translation into clinical setting to serve Veterans and Civilian survivors with SCI.

DETAILED DESCRIPTION:
Spinal cord epidural stimulation (ES) is a neuromodulation modality that can facilitate standing, stepping and walking with and without assistive devices in individuals with SCI, however; ES must be accompanied with locomotor training that at present requires a labor-intensive commitment from multiple well-trained personnel using specialized treadmill equipment. Exoskeletal assisted walking (EAW) on the other hand can be safely and efficiently used for ambulation after SCI in combination with ES without the use of other specialized equipment and multiple personnel. The investigators demonstrated that 12-weeks of EAW+ ES resulted in volitional stepping, with improved temporal and rhythmic electromyography (EMG) patterns and speed and with a reduction in EAW assistance to 35%. Unfortunately, EAW+ES does not appear to effectively restore lean mass below the level of injury, which impacts proprioceptive feedback to the spinal locomotor centers. Thus, in addition the investigators have demonstrated that 16-weeks of electrically-evoked resistance training (RT) resulted in robust muscle hypertrophy of the paralyzed knee and hip extensor muscle groups. Therefore, this proposal leverages these research programs by addressing two major gaps; 1) the use of combination EAW+ES as an activity-dependent plasticity tool for restoration of over ground locomotion and 2) enhancement of muscle quality using RT to provide afferent leverage for neuromodulation techniques.

Specific Aims:

1. To determine the impact of 12 months of EAW+ES+RT on 10-meter over ground walking-speed, number of EAW unassisted steps and EMG patterning compared to 12-months of EAW+ delayed-ES +no-RT (control group).
2. To determine the impact of 12-months of EAW+ES+RT on blood pressure, total and regional body composition, oxygen uptake as well as anabolic and inflammatory biomarkers compared to the control group.
3. To determine the impact of 12-months of EAW+ES+RT on parameters of bladder filling and emptying as measured by urodynamic studies compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. All participants will be between 18-60 years old, male or female, with traumatic motor complete SCI and level of injury of T10 and above, as determined by EMG testing and International Standards for Neurological Classification of SCI (ISNCSCI) exam.
2. Participants' knee extensors must respond to standard surface NMES procedures (frequency: 30 Hz; pulse duration:450 μs and amplitude of the current:200 mA) to ensure intact neural circuitry below the level of SCI.
3. All participants will undergo ISNCSCI examination for neurological level and function and only those with American Spinal Injury Classification (AIS A and B; i.e. motor deficit below the level of injury) will be included.

Exclusion Criteria:

1. Diagnosis of neurological injury other than SCI, including cauda equina or distal conus injuries resulting in limb or sacral areflexia;
2. Unhealed fracture in either lower or upper extremities;
3. Severe scoliosis, hip knee range of motion (ROM) or flexion knee contractures preventing positioning in an exoskeleton or plantarflexion contracture greater than 20 degrees.
4. Untreated or uncontrolled hypertension defined as high resting blood pressure greater than 140/90 mmHg and severe orthostatic hypotension (drop greater than 20 mmHg compared to resting supine blood pressure) or incapable to maintain a sitting or EAW standing posture;
5. Other medical conditions including cardiovascular disease, uncontrolled type II DM, uncontrolled hypertension, and those on insulin, pressures sores stage 3 or greater, or symptomatic urinary tract infection;
6. Unable to fit in the device for any reason;
7. Taking anti-coagulants or anti-platelet agents, including aspirin if unable to be off this medication for medical reasons;
8. Implanted pacemakers and/or implanted defibrillator devices;
9. DXA T-Score less than -2.5. Scans done will include total body, dual hips and knees. Total hip BMD T-scores < -3.5 and knee BMD scores of less than 0.6 g/cm2 68-71;
10. Functional upper and lower extremity ROM, strength, spasticity and skin integrity will also have assessed prior to enrollment in the program. The Modified Ashworth Scale will be used to ensure safety of the participants prior to engagement in the rehabilitation program. Participants with severe spasticity or limited ROM will be excluded from the trial. This is based on the Ekso® manufacturer's recommendations72;
11. Untreatable severe spasticity judged to be contraindicated by the site Physician;
12. Pressure ulcer of the trunk, pelvic area, or lower extremities of grade 3 or more;
13. Psychopathology documentation in the medical record or history that may conflict with study objectives;
14. Any condition that, in the judgment of the principal investigator or medical provider, precludes safe participation in the study and/or increases the risk of infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in 10-meter over ground walking-speed | Baseline to 12 months
  The investigators will measure the speed of walking and the time elapsed during 10 meter distance.
Change in EMG Pattern | Baseline to 12 months
  The investigators will record muscle activity from the major lower extremity muscle groups.

SECONDARY OUTCOMES:
Changes in Systolic and Diastolic Blood Pressure | Baseline to 12 months
  The investigators will measure resting and walking blood pressure on continuous basis
Changes in regional fat mass | Baseline to 12 months
  body composition will be measured using dual energy x-ray absorptiometry
Change in Oxygen uptake | baseline and every 6 months for 12 months
  measuring whole oxygen uptake during 6-minute walking test

OTHER OUTCOMES:
Changes in Bladder Filling and Emptying using Fluoroscopy and EMG | Baseline to 12 months
  The investigators will determine the impact of 12 months intervention on parameters of bladder filling and emptying as measured by urodynamic studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Gorgey, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorgey AS, Goldsmith J, Alazzam A, Trainer R. Effects of percutaneously-implanted epidural stimulation on cardiovascular autonomic function and spasticity after complete spinal cord injury: A case report. Front Neurosci. 2023 Feb 16;17:1112853. doi: 10.3389/fnins.2023.1112853. eCollection 2023. PMID 36875669